CLINICAL TRIAL: NCT00175604
Title: Comparative Trial of Botox Versus Conventional Treatment Used in the Management of Children With Congenital Muscular Torticollis (CMT)
Brief Title: Comparative Trial of Botox in the Management of Children With Congenital Muscular Torticollis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Not able to recruit any subjects for the study and was closed in February 2008
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Stephen Tredwell, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C03-0550; W03-0164
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2011-02

CONDITIONS: Torticollis
Keywords: Botox; torticollis; Congenital Muscular Torticollis (CMT)
MeSH Terms: conditions — Torticollis; Congenital torticollis | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Botox — The babies that require a neck collar for CMT will be randomly placed into two groups. One group will receive standard treatment which includes physiotherapy and occupational therapy. The other group will receive standard treatment plus an injection of Botox.

SUMMARY:
The primary purpose is to investigate the effect of Botox on the treatment of congenital muscular torticollis (CMT). The investigators' hypothesis is that a Botox injection will be an effective treatment when used in conjunction with current treatment procedures.

DETAILED DESCRIPTION:
The babies that require a neck collar for CMT will be randomly placed into two groups. One group will receive standard treatment which includes physiotherapy and occupational therapy. The other group will receive standard treatment plus an injection of Botox. The babies will be monitored to determine if one group has a more favorable outcome than the other in terms of range of motion, length of treatment time and number of required surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Infants diagnosed with CMT and referred by family physician, pediatrician or orthopaedic surgeon
* Initial assessment and initiation of treatment prior to 4 months of age
* Cervical spine radiograph, no focal bony abnormality
* Head tilt greater than 5 degrees at 5 months of age
* Lateral head righting past neutral in upright suspension
* Restricted neck range of movement in lateral flexion or rotation or both
* Signed consent form and willingness to participate in the study
* Compliance with attending bi-weekly follow-up appointments

Exclusion Criteria:

* Any other diagnosis affecting tone or muscle function
* Any condition that would preclude an anesthetic
* Any vertebral abnormalities identified by radiograph
* Attending other health practitioners for treatment, i.e., massage therapist, chiropractor
* Any associated ocular problems as determined by a pediatric ophthalmologist

Ages: 4 Months to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2004-08; Primary Completion 2008-02 (Estimated); Study Completion 2008-02 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be range of motion. | assessed bi-weekly until treatment is complete

SECONDARY OUTCOMES:
The secondary outcomes will be length of treatment time and number of required surgeries. | assessed bi-weekly until treatment is complete

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Tredwell, MD, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Children's Hospital, Dept. of Orthopedics, Vancouver, British Columbia, Canada